CLINICAL TRIAL: NCT01886833
Title: An Observational Study to Evaluate Causes of Rotavirus Vaccine Failure in Zambian Children in the Context of Routine Immunization Services
Brief Title: Causes of Rotavirus Vaccine Failure in Zambian Children
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Roma Chilengi, Dr, Centre for Infectious Disease Research in Zambia
Other Study IDs: ROVAS 01; 1R01AI099601-01 (NIH)
Record Dates: First submitted 2013-06-22; First posted 2013-06-26 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Diarrhoea
Keywords: Rotavirus; Diarrhoea; Immunisation; Seroconversion; Breastmilk; HIV; Zinc; Vitamin A; Failure
MeSH Terms: conditions — Diarrhea; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for immunogenicity testing will be analyzed in batches.
  Stool samples for rotavirus extraction will also be stored and analyzed in batches.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mother-Infant Pair: The study will involve consenting mother-infant pairs from Kamwala health facility in Lusaka where the Maternal Child Health (MCH). Those generally interested will be invited to the research clinic, where more detailed information about the study is offered. Motivated mothers will be recruited and taken through the written informed consent process by the study nurse.
  Enrolled mother-infant pairs will undergo baseline procedures as earlier described. They will then be followed prospectively until about December 2016. They will be expected to come to the clinic for scheduled visits at baseline, 1, 3, 12, 15 and 42 months. They will be urged to come to the clinic for unscheduled visit should the infant be unwell at any time, and particularly each time the infant experiences diarrhoea.

SUMMARY:
Zambia recently introduced routine infant immunization against rotavirus - the most important cause of severe gastroenteritis and diarrhoea mortality in children. Although vaccines like Rotarix are a cost effective tool against infectious diseases, live oral vaccines can be less immunogenic and efficacious in developing world settings as compared with industrialized countries. Reasons behind this phenomenon are not well understood, but may relate to continued maternal antigen exposure and high level maternal immunity that is passed to the foetus/newborn transplacentally and/or through breast milk.

Therefore, three arising hypotheses include: (i) high-level rotavirus-specific maternal immunity (in the form of anti-rotavirus breast-milk immunoglobulin A (IgA) and transplacental serum IgG) is a major contributor to failed seroconversion following infant vaccination. (ii) Malnutrition negatively impacts infant immunity and increases the risk of post-vaccination rotavirus gastroenteritis. (iii) Introduction of rotavirus vaccine will alter the molecular epidemiology of circulating rotavirus strains detected in vaccinated children presenting with severe diarrhea.

To address these hypotheses, the proposed study will recruit a prospective cohort of 420 mother-infant pairs. These will be enrolled at the time of vaccination and followed for up to four years. Baseline immunological status will be ascertained and seroconversion rates determined a month after full immunization. Incident rotavirus gastroenteritis will be monitored in the vaccinated infants whenever episodes of diarrhoea occur; through this surveillance, the sero-strains of rotaviruses causing disease will be tracked over the four year period. Contributions of HIV infection both in mothers and infants, vitamin A and zinc deficiency, weight for age Z-scores as well as mid upper arm circumference will also be assessed. Knowledge gained from this study will inform future interventional trials on strategies to improve rotavirus vaccine effectiveness in the developing world.

DETAILED DESCRIPTION:
The study will be conducted at Kamwala health facility in Lusaka where the Maternal Child Health (MCH) and antiretroviral therapy (ART) clinics as well as the Centre for Infectious Disease Research Zambia (CIDRZ) Kamwala Research Unit are co-located. Kamwala has a catchment population of over 10,000 with approximately 30 new infants presenting to MCH each month with 6-14 week (DPT-HiB-Hep) immunisation rates above 95%. Mother-infant pairs will be approached during the initial visit to MCH by the study clinic assistant or peer counsellor with information about this study in the local language of choice. Those generally interested will be invited to the research clinic which is close by, for more detailed information during which motivated mothers will be recruited and taken through the written informed consent process by the study nurse. For illiterate participants, an independent, literate individual will witness and validate the informed consent process. A specific log will be maintained to show information on dates and numbers of those invited to the study, reasons for refusal documented.

A senior research nurse, study nurse, and clinical research assistant will be responsible for informed consent and enrolment procedures under the supervision of the investigator. A paediatrician will be available for hands-on consultation when needed.

Cohort Follow-up. Enrolled mothers will be asked to complete demographic and behavioural questionnaires, a participant locator form, and undergo phlebotomy and mechanical expression of breast-milk at the enrolment visit for determination of anti-rotavirus IgG and IgA (in serum and breast-milk). Infants will have a baseline anti-rotavirus IgA and IgG antibodies determined to ascertain baseline exposure to wild-type and transplacental immunoglobulin followed by a second serum IgA determination one month following completion of rotavirus vaccination (at approximately 14-20 weeks).

Infants will then be followed quarterly in-clinic for the remainder of the study and will also make interim clinic visits if the child has diarrhoea. At each visit, the child will be weighed, height measured, and anthropometrics taken, including skin fold for subcutaneous body fat and mid upper arm circumference. During any symptomatic interim visits, assessments will be made of disease severity (by Vesikari scale) and a sample of stool will be collected for determination of rotavirus antigen and genotype if rotavirus positive. The patient will also be sent home with a diarrhoea diary to be completed over the following two weeks. Following identification of an child with severe gastroenteritis, an age-matched control from within the cohort (without recent gastroenteritis) will be brought in for measurement of Vitamin A and serum zinc levels. Children with gastroenteritis will be treated according to national guidelines (per World Health Organization (WHO) Integrated Management of Childhood Illness). If referral is required, the child will be referred to outpatient clinic, or in serious cases the University Teaching Hospital.

Study Procedures. Same as above.

Laboratory Methods.

1. Detection of Rotavirus-specific IgA and IgG will occur by ELISA. Detection of rotavirus-specific IgA and IgG will occur by ELISA. Briefly, the procedure is as follows. Microplate wells (e.g., Nunc Immuno I) are incubated with purified viral antigen preparations, then washed with phosphate buffered saline with Tween detergent (PBS-T). Serum and breast-milk samples are diluted serially (in PBS-T containing 1% bovine serum albumin) and incubated in the coated microplates for 2 hours at 37oC then overnight at 4oC. Microplates are then washed and peroxidase-conjugated anti-human IgA or IgG goat antibodies (Sigma Immunochemicals) is added. The reaction is then terminated with H2SO4, and optical density is measured by EIA plate reader. All samples are assayed in duplicate against each viral antigen and against a control antigen. A test well was considered positive by its optical density at 450 nm, e.g., if it is greater than or equal to two times that of its own control. Specificity is controlled by including wells containing control antigen incubated in the absence of the sample, and sensitivity is checked by including wells containing viral antigen incubated in the presence of samples known to contain high titre of a particular rotavirus-specific immunoglobulin class.
2. Detection of Rotavirus Antigen will occur by Rotaclone ELISA. Stool samples will be tested for rotavirus by ELISA (Rotaclone®, Meridian Biosciences) according to manufacturer's specifications. Briefly, sample will be brought to room temperature and diluted with buffered saline with 0.02% thimerosol. Diluted sample and enzyme conjugate are then incubated with a monoclonal antibody to the VP6 protein within the Rotaclone microplate. Substrate buffers containing urea peroxide and tetramethylbenzidine are then added, and the reaction is terminated with H2SO4. Spectrophotometric determination of result is then made by measuring absorbance at 450 nm against an air blank. Specimens with absorbance units (A450) greater than 0.150 are considered positive. Those with absorbance equal to or below 0.150 are considered negative.

3 Determination of Rotavirus VP7 Genotype. Viral RNA is extracted from a 10% suspension of rotavirus antigen-positive faecal material in PBS (pH 7.0) using TRIzolTM Reagent (GIBCO Life Technologies) according to the manufacturer's protocol. Viral RNA is then taken through RT-PCR as described earlier.

Extracted viral RNA is then taken through nested PCR utilizing primers which are complimentary to the 3' ends of both viral RNA strands within gene segment 9, which encodes viral protein 7 (VP7). These primers are used for first strand synthesis. Primer RVG9 and six serotype-specific primers (aBT1, aCT2, aET3, aDT4, aAT8, and aFT9) which are located in six variable regions on the gene 9 and correspond to G-serotypes 1, 2, 3, 4, 8 and 9, are used in second amplification. Briefly, 5 µl of RNA with 25 pmol of each primer Beg9 and End9 is denatured for 5 min at 97°C and cooled on ice. Thereafter, 8 µl of RT reaction mixture containing 1.5 µl of 10X PCR buffer (500 mM KCl, 100 mM Tris-HCl (pH 8.3), 2 µl of 25 mM MgCl2, 2 µl of 2.5 mM of each dATP, dCTP, dGTP and dTTP, 10 U AMV reverse transcriptase (Promega) and 20 U Rnasin ribonuclease inhibitor (Promega), is added to the sample-primer mixture and incubated at 42°C for 60 min. PCR buffer mixture (35 µl), containing 3.5 µl of 10X PCR buffer, 2 µl of 2.5 mM peach dATP, dCTP, dGTP and dTTP, 2.5 U AmpliTaq DNA polymerase (Perkin Elmer) and 27 µl of water are added to RT reaction. The reaction mixture is denatured at 94°C for 3 min, followed by 30 cycles (1 min at 94°C, 2 min at 42°C, 3 min at 72°C) and a final extension of 5 min at 72°C.

First-round PCR products (2 µl) are transferred to 48 µl of second PCR reaction mixture, containing 5 µl of 10X PCR buffer, 25 pmol each primers aBT1, aCT2, aET3, aDT4, aAT8, aFT9 and RVG9, 0.2 mM each dATP, dGTP, dCTP and dTTP, 2mM MgCl2, 2.5 U of Taq polymerase. Second-round cycling conditions are identical to first round, except that only 25 cycles are run. The PCR products are analyzed by gel electrophoresis to identify expected lengths of amplified VP7, allowing determination of genotype. Other primer sets, PCR conditions and/or sequencing is used to distinguish genotype when/if the initial primers fail.

4 Determination of VP4 Genotype. The strategy for PCR typing of gene 4 is identical, in principle, to that used for VP7.64 First strand synthesis (reverse transcription) takes advantage of highly conserved areas of VP4 utilizing primers Con2 and Con3 (Box 3), which are complimentary to the 3' ends of both viral RNA strands within gene segment 4. 1 to 5 µL of viral RNA is added to 0.5 ml microcentrifuge tubes containing 3.5 µl of dimethylsulfoxide (Sigma) in a final volume of 8.5 µl, and the samples are mixed and denatured at 97°C for 5 min. The samples are then cooled on ice for 5 min and collected by brief centrifugation. 13.5 µL of H20, 16 µL of deoxynucleoside triphosphates (1.25 mM each dATP, dGTP, dCTP, and dTTP), 5 µL 1OX buffer (100 mM Tris-hydrochloride [pH 8.3], 500 mM KCl) (Perkin-Elmer Cetus), 3.5 µL of 25 mM MgCl2, 2 µl of primer (containing 25 µM of each primer, Con 2 and Con 3), and 9 U reverse transcriptase is then added to each denatured dsRNA sample tube (to give a final reaction volume of 49 µ1) and incubated at 42oC for 60 minutes.

Following addition of 1 µL (1.9U) of Taq polymerase and 100 µL mineral oil, first-round PCR is carried out for 30 cycles (1 min 94oC, 2 min at 50oC, and 2 min at 72oC. A cooling cycle is used to bring the samples to 17OC at the completion of the experiment. The second-round typing reaction if performed using 0.5 to 5 µL of the first-round product (5 µL if no visible product; 0.5 µL if visible product) is mixed with 45 µL reaction mixture in a final volume of 50 µL. If less than 5 µL of first round product is added, the remaining volume, to complete 50 µL, is 10mM TrisHCl (pH 8.3)-2.5mM MgCl¬2. The reaction mixture is 19.5 µL water, 16 µL dNTPs, 5 µL 10X Buffer II, 3 µL 25 mM MgCl2, 1 µL of the primer cocktail (containing 20 µM each of Con3, 1T-1, 2T-1, 3T-1, and 4T-1), and 0.5 µL (2.5U) Taq. The samples are overlaid with mineral oil and taken through 25 rounds of PCR (same cycles as first round). The samples are then analyzed by gel electrophoresis and product size enables determination of VP4 genotype. Other primer sets and/or sequencing is used to distinguish genotype when/if the initial primers fail.

5 Determination of Vitamin A and Zinc levels: Serum samples will be evaluated for Vitamin A level by ELISA (e.g., Human Vitamin A, EIAAB) according to the manufacturer's instructions. Briefly, the microtitre plate provided in this kit has been pre-coated with an antibody specific to Vitamin A. Standards or samples are then added to the appropriate microtitre plate wells with a biotin-conjugated polyclonal antibody preparation specific for VA and Avidin conjugated to Horseradish Peroxidase (HRP) is added to each microplate well and incubated. Then a tetramethylbenzidine substrate solution is added to each well. Only those wells that contain Vitamin A, biotin-conjugated antibody and enzyme-conjugated Avidin will exhibit a change in colour. The enzyme-substrate reaction is terminated by the addition of a H2SO4 and the color change is measured spectrophotometrically at a wavelength of 450 nm. The concentration of VA in the samples is then determined by comparing the O.D. of the samples to the standard curve.

Zinc levels will be measured from blood using assays such as Lampugnani's simple colorimetric method which uses a spectrophotometric method with chromogen 4-(2-pyridylazo) resorcinol sodium salt to measure serum zinc concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Mother willing to participate voluntarily and able to provide signed informed consent (with witness in the case of illiterate participant)
* Infant eligible for rotavirus vaccine immunization as per national policy (male or female infant, 6-12 weeks old)
* Mother willing to undergo study procedures, including questionnaires, HIV counselling and testing, CD4 testing, and provide breast milk and blood sample at enrolment.
* Mother willing for child to undergo study procedures including full-course rotavirus vaccination, phlebotomy at enrolment and 1 month post-rotavirus vaccination, and presentation to clinic for collection of stool sample when infant has diarrhoea.
* Plans to remain resident in the area and willing to come for scheduled visits for the duration of the study.

Exclusion Criteria:

* Contraindication to rotavirus vaccination.
* Previous administration of rotavirus vaccine to child.
* Recent immunosuppressive therapy in child (including high-dose systemic corticosteroids).
* History of ever receiving a blood transfusion or blood products, including immunoglobulins within the last 6 months, for mother and child.
* Mother plans for herself or child to move away from the study catchment area within the next two years.
* Any condition deemed by the study investigator to pose potential harm to the participants or jeopardize the validity of study results.

Ages: 6 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother-infant pairs presenting for MCH at Kamwala health facility in Lusaka and where the infant is 6-15 weeks old, will be recruited into the cohort and followed for a period of 1-4 years depending on time of enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, MD, MSc, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 420 mother-infant pairs were recruited between April 2013-March 2014 from Kamwala Health Care Clinic during routine immunisation. Enrolled mother-infant pairs will undergo baseline procedures and were followed prospectively until March 2017 at scheduled visits at baseline, 1, 3, 12, 15 and 42 months. and unscheduled visits if infant was unwell.
Groups:
- Mother-infant Pair IgA: Proportion of Immunized Infants Exposed to High Breast Milk anti-rotavirus IgA Who Fail to Seroconvert will be calculated comparing baseline to after 1 month of full immunization.
Period: Overall Study
Arm/Group | Mother-infant Pair IgA
Started | 420
Completed | 216
Not Completed | 204
Not completed — IgA not available from both periods | 204

BASELINE CHARACTERISTICS:
Arm/Group | Mother-Infant Pair
Number analyzed (Participants) | 420
Age, Continuous [Mean (Full Range); unit: months] | 27 [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232
  Male | 188
Region of Enrollment [Number; unit: participants]
  Zambia | 420

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Immunized Infants Exposed to High Breast Milk Anti-rotavirus Immunoglobulin-A Who Fail to Seroconvert
Description: The primary exposure in this cohort is maternal IgA status, as we believe breast milk IgA is the most critical factor in failed vaccination, and maternal IgA has previously been estimated to be either high level (approximately 55%) or undetectable or low level (approximately 45%).
  We will collect maternal serum and breast-milk IgA at the time of vaccination and then measure infant anti-rotavirus-specific serum IgA levels 1 month following the second dose of Rotarix™ (GlaxoSmithKline) rotavirus vaccine.
Time Frame: 1 month following full immunization
Population: Of the 420 participants that were enrolled in the study, we had rotavirus specific paired IgA at baseline and post vaccination for 216 infants.
Measure: Number; unit: Proportion of exposed infants
Groups:
- Mother-Infant Pair: The proposed study will recruit a prospective cohort of 420 mother-infant pairs. These will be enrolled at the time of vaccination (6-12 week old infant) and followed for up to four years. Baseline immunological status will be ascertained and seroconversion rates determined a month after full immunization.
Arm/Group | Mother-Infant Pair
Number analyzed (Participants) | 216
Proportion of exposed infants | 0.602

2. Primary Outcome: Proportion of Immunized Infants Exposed to Transplacentally-acquired, Rotavirus-specific, Infant Serum IgG Who Fail to Sero-convert.
Description: The co-primary exposure in this cohort is transplacentally acquired anti-rotavirus immunoglobulin-G.
  We will collect infant serum at baseline before any vaccination and then measure the levels of anti-rotavirus-specific serum IgG and will also obtain the same at 1 month following the second dose of Rotarix™ rotavirus vaccine.
Time Frame: 1 month after full immunisation
Population: We did not test the serum IgG collected at 1 month following the second dose of Rotarix™ rotavirus vaccine because all infants were seropositve at baseline
Arm/Group | Mother-Infant Pair
Number analyzed (Participants) | 0

3. Primary Outcome: Proportion of Immunized Infants Exposed to Maternal HIV Infection Who Fail to Seroconvert
Description: To evaluate whether maternal HIV infection (as well as level of CD4 count) affects infant vaccine take, we will collect the maternal HIV status, (and CD4 count if +ve). We will then correlate the maternal HIC status and CD4 count levels to infant zero conversion at 1 month after the two vaccine doses.
Time Frame: 1 month after the two vaccine doses
Population: Of the 420 mothers, 125 were confimed HIV+
Measure: Number; unit: Proportion of exposed infants
Groups:
- Mother/Infant Pair: The proposed study will recruit a prospective cohort of 420 mother-infant pairs. These will be enrolled at the time of vaccination (6-12 week old infant) and followed for up to four years. Baseline immunological status will be ascertained and seroconversion rates determined a month after full immunization.
Arm/Group | Mother/Infant Pair
Number analyzed (Participants) | 125
Proportion of exposed infants | 0.704

4. Secondary Outcome: Proportion of Immunized Infants With Low Micronutrient Levels (as Indicated by Serum Zinc and Vitamin A), Who Fail to Seroconvert
Description: To evaluation whether nutritional status affects vaccine take, we will assess the immunized infant's nutritional status as indicated by serum level of zinc and vitamin A. These will be correlated to seroconversion results.
Time Frame: 1 month after full immunization
Population: Of the 216 infants with paired serum IgA at baseline and after 1 month of complete immunization, 164 had deficient micronutrients
Measure: Number; unit: Proportion micronutritionally deficient
Arm/Group | Mother-Infant Pair
Number analyzed (Participants) | 164
Proportion micronutritionally deficient | 0.5

5. Other Pre Specified Outcome: Sero-epidemiology of Breakthrough Rotavirus Infection in Immunized Infants
Description: Determination of genotype in every rotavirus causing severe gastroenteritis will be done each time stool samples are collected for diarrhoea. Patients presenting with any diarrhoea will be tested for rotavirus and staged clinically (by Vesikari score). Those with severe disease (e.g., Vesikari >11/20) will be processed for genotype. Thus, we will identify the number of rotavirus cases following vaccination as well as identify the strain in those with severe disease.
  This will allow for "wild type versus vaccine"strain mismatch evaluation. We anticipate that the circulating strains in the community will change in response to vaccine pressure at the population level. However, when interpreting reasons for vaccine failure, it is critically important to evaluate strain mismatch because the way to approach this type of breakthrough disease is dramatically different than if there is breakthrough infection to vaccine strain rotavirus.
Time Frame: 42 months
Population: There were 81 episodes of diarrhoea from which samples were collected. 15 were positive for rotavirus by EIA
Measure: Count of Units; unit: stool samples
Units Other Than Participants: stool samples
Groups:
- Infants: Determination of genotype in every rotavirus causing severe gastroenteritis will be done each time stool samples are collected for diarrhoea. Patients presenting with any diarrhoea will be tested for rotavirus and staged clinically (by Vesikari score). Those with severe disease (e.g., Vesikari >11/20) will be processed for genotype. Thus, we will identify the number of rotavirus cases following vaccination as well as identify the strain in those with severe disease.
Arm/Group | Infants
Number analyzed (Participants) | 81
Number analyzed (stool samples) | 81
stool samples
  G1P8 | 4
  G2P6 | 3
  G1P6 | 2
  Untypable | 6
  Negative for rotavirus | 66

ADVERSE EVENTS:
Time Frame: 4 years
Description: The quarterly in-clinic follow up of infants will invariably lead to early identification of medical problems. These will be treated immediately in the clinic as per national guidelines. Cases needing hospitalization will be transferred to the University Teaching Hospital.
Arm/Group | Mother-Infant Pair
Serious Adverse Events (participants affected / at risk) | 51/420
Other Adverse Events (participants affected / at risk) | 0/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mother-Infant Pair (N=420)
fever and convulsions (General disorders) | 2 (2) — fever and convulsions prior to death
Hospitalization (General disorders) | 39 (39) — 39 children were hospitalized with various conditions not related to the study
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Diarrhoea followed by death
Diarrhoea plus vomiting (Gastrointestinal disorders) | 1 (1) — Diarrhoea plus vomiting followed by death
acute pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — acute pneumonia followed by death
severe burns (Social circumstances) | 1 (1) — severe burns followed by death
Fever and malaria (Infections and infestations) | 1 (1) — Fever and malaria followed by death
injuries (Injury, poisoning and procedural complications) | 1 (1) — injuries from road traffic accident followed by death
death from unknown causes (General disorders) | 4 (4) — Death from unknown causes

LIMITATIONS AND CAVEATS:
If vaccine strains are a mis-match of vaccine strain and non-vaccine strain that remains constant and unchanged over time, it would favour multiple reasons for vaccine failure, making identification of solutions difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No